CLINICAL TRIAL: NCT00354965
Title: A Study to Determine PK Profiles of AUGMENTIN XR in Adolescents Weight at Least 40 kg Receiving Augmentin XR BID for 10 Days
Brief Title: Pharmacokinetic Profiles Of Amoxicillin 2000 mg And Clavulanate 125 mg In Adolescent Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUG102821
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Infections, Respiratory Tract
Keywords: ABS; Acute Bacterial; Sinusitis; Bacterial Sinusitis
MeSH Terms: conditions — Respiratory Tract Infections; Sinusitis | interventions — Amoxicillin-Potassium Clavulanate Combination

ARMS (1):
- ARM 1 (Experimental)
  Interventions: Drug: amoxicillin/clavulanate potassium

INTERVENTIONS:
Drug: amoxicillin/clavulanate potassium — amoxicillin/clavulanate potassium

SUMMARY:
Clinical research study to test amoxicillin and clavulanate tablet formulation for use in Acute Bacterial Sinusitis (ABS) in adolescent patients weighing at least 40 kilogram (kg) and no more than 16 years old. ABS is an acute bacterial infection of the sinus. The purpose of this study is to find out how children tolerate Augmentin XR and what happens to Augmentin XR in the body after it has been swallowed by children.

ELIGIBILITY:
Inclusion criteria:

* Patient weighs at least 40 kg.
* Younger than 16 years old (no older than their 16th birthday).
* Suspected acute bacterial sinusitis.
* Able to swallow amoxicillin/clavulanate tablets.

Exclusion criteria:

* Personal or family history of adverse reactions or hypersensitivity or allergy to any penicillin or cephalosporin antibiotics.
* History of reaction to multiple allergens (if considered clinically relevant by the principal investigator).
* Patient is participating in another clinical trial or has received or anticipates receiving an investigational drug, vaccine, or medical device prior to the first dose of study medication or during the conduct of the study.
* History or presence of gastrointestinal, hepatic or renal disease or other conditions known to or that may interfere with the absorption, distribution, metabolism or excretion of study medication.
* Treatment with probenecid or allopurinol within 7 days of study entry.
* Female patients with a positive urine hCG (human chorionic gonadotropin) test at screening, or who are lactating (breast feeding) or are unwilling to be abstinent until completion of the follow-up visit.
* History of diarrhea due to Clostridium difficile following treatment with antibiotics.
* History of hypersensitivity or allergy to heparin or related preparations (if the clinical research unit uses heparin to maintain intravenous cannula patency).
* Patient is diagnosed with mononucleosis.
* Estimated Glomerular Filtration Rate (GFR) <40 ml/min.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2006-01-19 (Actual); Primary Completion 2007-04-02 (Actual); Study Completion 2007-04-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic data on amoxicillin/clavulanate | Time above MIC (T>MIC)for amoxicillin when amoxicillin/clavulanate is given orally twice daily to adolescents.

SECONDARY OUTCOMES:
Safety, tolerability, and clinical response of oral amoxicillin/clavulanate | twice daily for 10 days in adolescent patients.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Sylva, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Erie, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study AUG102821 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/AUG102821?search=study&search_terms=AUG102821#rs
- Available data/document: Dataset Specification: AUG102821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AUG102821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AUG102821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AUG102821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AUG102821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AUG102821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register